CLINICAL TRIAL: NCT06368947
Title: Therapeutic Play on Pain Tolerance and Emotion Regulation in Children Receiving Chemotherapy
Brief Title: Therapeutic Play on Pain Tolerance and Emotion Regulation in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ARZU SARIALİOĞLU, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/172
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Play Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Therapeutic play sessions will be organized twice a week for 4 weeks during chemotherapy treatment for children diagnosed with acute lymphoblastic leukemia in the intervention group.
  Interventions: Behavioral: Therapeutic Play
- control (No Intervention): Routine treatment will be applied to children in the control group receiving chemotherapy during their treatment.

INTERVENTIONS:
Behavioral: Therapeutic Play — Therapeutic play sessions will be organized twice a week for 4 weeks during chemotherapy treatment for children diagnosed with acute lymphoblastic leukemia in the intervention group.
  Arms: intervention

SUMMARY:
The research is a randomized controlled experimental study. The population of the research will consist of 10-18 year old children who were diagnosed with acute lymphoblastic leukemia and received chemotherapy, who were admitted to the Children's Hematology Clinic of Adana City Training and Research Hospital between 19.05.2024 and 19.05.2025. Therapeutic play sessions will occur over a 4-week period during chemotherapy treatment.

DETAILED DESCRIPTION:
Type of Research: The research is a randomized controlled experimental study. Place and Time of the Research: The research will be carried out at the Pediatric Hematology Clinic of Adana City Training and Research Hospital between April 2024 and June 2026.

Population and Sample of the Research: The population of the research will consist of 10-18 year old children who were diagnosed with acute lymphoblastic leukemia and received chemotherapy, who were admitted to the Children's Hematology Clinic of Adana City Training and Research Hospital between 19.05.2024 and 19.05.2025. In this study, G-power prior power analysis was performed to determine the sample size. In the power analysis, it was determined that if the study was conducted with a total of 60 participants in two groups with 30 participants in each group for the t test in independent groups, 80% power could be achieved with a 95% confidence interval at a significance level of 0.05. It was decided to collect data from a total of 66 children by including a 10% backup sample in this number in case of data loss.

Therapeutic game: In the research, a preliminary application will be made first. A special play bag will be created for each child patient, which will not threaten his health and can be disinfected. Therapeutic play sessions will occur over a 4-week period during chemotherapy treatment. Therapeutic game 2 days a week for a maximum of 60 minutes. It will be carried out for 4 weeks.

Week 1: It will consist of meeting, building trust, giving information about the sessions, and planning the therapeutic game. After the initial meeting and trust building stages, activities will be held with emotion cards. Week 2: The researcher will carry out activities that will enable the child to express his emotions through puppet making. A puppet with the characteristics desired by the child will be made by the child and the researcher. The shape and appearance of the puppet will be determined by the child.

Week 3: At this stage, after the puppet is completed, the drama will be created and realized through the meaning given to the puppet and the emotions reflected. Emotions will be discussed on the puppet, and the child will be helped to understand, express and analyze his feelings.

Week 4: The child and the researcher will produce creative stories and the child's emotions will be discussed. In the last sessions of this stage, the child will be comforted by using the "healing stories for children" book.

Evaluation of Data The data will be analyzed with the SPSS for Windows 22 package program. The normality distribution of the data will be determined by Kurtosis and Skewness coefficients. In the analysis of the data, in addition to numbers, percentages, averages and standard deviations, t-test will be used in independent groups for normally distributed measurements and Mann Whitney U analysis will be used for non-normally distributed measurements in comparing paired groups. Statistical significance will be accepted as p<0.05.

Ethical Principles of Research In order to conduct the research, official permission was obtained from the relevant institution with ethical approval from the Ataturk University Non-Interventional Clinical Research Ethics Committee. Clinical trials will be registered for randomized controlled studies. The purpose of the study will be explained to children and parents who meet the research group criteria, their questions will be answered, and their verbal and written consent will be obtained. Children and parents will be informed that the data collected during the research will be processed confidentially and anonymously, will not be used outside of the study in question, and that they can leave the study at any time. Since the research is based on the use of data obtained from humans, and therefore the need to respect personal rights, the relevant ethical principles of "Informed Consent", "Volunteering" and "Protection of Confidentiality" will be followed. The "Principle of Equality" will be tried to be fulfilled by giving the children in the control group the same game bags given to the children in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 10-18
* Diagnosed with acute lymphoblastic leukemia
* Those receiving chemotherapy treatment
* Children who do not have a chronic disease other than the diagnosis of the disease in question

Exclusion Criteria:

* Under 10 years of age or over 18 years of age
* Diagnosed other than acute lymphoblastic leukemia
* Not receiving chemotherapy treatment
* Children with chronic diseases other than the diagnosis of the disease in question

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-12-29 (Actual); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
Pain Tolerance Scale for Children with Cancer | 12 months
  The scale was created to develop a tool to measure psychological acceptance in children experiencing pain during cancer treatment. The test version of the scale was conducted on children between the ages of 7 and 18 who were receiving cancer treatment. The Turkish reliability and validity study of the scale was conducted and it was found suitable for use in Turkish children with cancer. The scale is a 7-point Likert type scale consisting of 20 items (0 = strongly disagree and 6 = strongly agree). Some items in the scale (1, 2, 3, 5, 6, 7, 8, 9, 11, 13, 14, 15, 16, 18, 20 items) are reverse coded. The minimum score to be obtained from the scale is 0 and the maximum score is 120. Increasing scale scores indicate an increase in the level of acceptance.
Emotion Regulation Scale for Children and Adolescents | 12 months
  The scale was adapted to Turkish in 2021. The scale is a self-rating scale created to evaluate the differences in the use of two emotion regulation strategies. The scale consists of two subscales, reappraisal and suppression, and 10 items. Evaluation is made with a 5-point Likert type rating. Items 1, 3, 5, 7, 8, and 10 of the reevaluation subscale; Items 2, 4, 6, and 9 represent the suppression subscale. High scores obtained from the subscales indicate that the emotion regulation strategy represented by the subscale is frequently used.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University Nursing of Faculty, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
THE ARTICLE IS INTENDED TO BE SHARED AFTER IT IS PUBLISHED